CLINICAL TRIAL: NCT05507788
Title: Wheelchair Seating: An Assessment of Multicell Air Cushions on Sitting Posture and Limits of Stability
Brief Title: Multicell Air Cushions: Sitting Posture and Limits of Stability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Jonkoping University (Other)
Responsible Party: Principal Investigator, David Rusaw, Associate Professor, Jonkoping University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETAC
Record Dates: First submitted 2022-04-28; First posted 2022-08-19 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Wheelchairs; Self-Help Devices; Posture; Sitting Position; Limits of Stability; Balance

STUDY DESIGN:
Intervention Model Description: The convenience sample of 15 individuals will each complete the test protocol under the 3 seating conditions in random order.
Masking Description: Efforts will be taken to mask the conditions to the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cushion (Experimental): Three seating conditons (Quadtro Select 10cm, Starlock 10cm, and Starlock 13cm)
  Interventions: Device: Wheelchair air cushion

INTERVENTIONS:
Device: Wheelchair air cushion — Reaching tasks during each of the seating conditions decribed in the Arms section.

SUMMARY:
The study's aim is to assess the sitting and dynamic postural control of stability of wheelchair users who have compromised postural control and risk of ulcers while using individually adjusted multi-cell air cushions with and without individual cell-locking function and variable depths.

ELIGIBILITY:
Inclusion Criteria:

* individuals who use a wheelchair
* have used a wheelchair for no less than 2 years
* score from 3-6 on the Functional Independence Measure
* not currently inpatients or those currently accessing acute care for concomitant health-related issues

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Reach distance | Day 1
  the linear distance from the start position to the furthest reach point during the trial
Accuracy | Day 1
  the ratio of the minimum distance (straight line) from the start position to the total distance traveled until the furthest reach point
Time | Day 1
  length of time from the start position to furthest reached point
total path length of Center of Pressure | Day 1
mean velocity of Center of Pressure | Day 1
pressure-distribution between the seating surface and the two foot Force-sensing arrays | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: David F Rusaw, PhD, Principal Investigator — Jonkoping University
Locations (1):
- Jönköping University, Jönköping, Sweden

IPD SHARING:
Plan to Share IPD: No